CLINICAL TRIAL: NCT05778214
Title: A Multi-Center, Randomized, Non-Inferiority, Prospective and Parallel-Group Trial to Evaluate the Safety and Efficacy of the Interventional Robotic System for Cerebral Angiography
Brief Title: A Clinical Trial for the Interventional Robotic System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Dean of the Department of Neurosurgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P01-QR-003
Record Dates: First submitted 2023-02-23; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Angiography
Keywords: Cerebral Angiography; Interventional Surgical Robot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Robotic System Assisted Surgery (Experimental): Experimental group underwent cerebral angiography using the vascular interventional surgical control system
  Interventions: Device: Interventional Robotic System
- Traditional Manual Surgery (No Intervention): The control group process the traditional manual operation for cerebral angiography

INTERVENTIONS:
Device: Interventional Robotic System — Cerebral angiography was performed by using the interventional robotic system
  Arms: Interventional Robotic System Assisted Surgery

SUMMARY:
The goal of this multi-center clinical trial is to evaluate the efficacy and safety of the interventional robotic system for cerebral angiography, researchers will compare the ordinary angiography to assess the clinical success rate, operation time, radiation absorption, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 85 years;
2. Plan to undergo cerebral angiography;
3. Voluntarily participated in this trial and signed the informed consent form.

Exclusion Criteria:

1. Preoperative mRS score >2;
2. Allergy or intolerance to iodine contrast media;
3. Allergy to interventional devices;
4. Severe cardiac, hepatic and renal insufficiency;
5. Active systemic infection;
6. Severe stenosis, occlusion or skin infection at the puncture site;
7. Subjects who are to undergo surgery at the same time as cerebral angiography;
8. Subjects with severe coagulation disorders, bleeding tendencies, or contraindications to anticoagulant drugs (e.g., heparin);
9. Subjects who are enrolled in clinical studies with other devices or drugs 3 months prior to screening;
10. Female subjects of childbearing age who are pregnant or breastfeeding;
11. Other subjects who, in the judgment of the investigator, are not suitable for participation in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Rate | at the end of surgery
  Assessment of the clinical success rate of the surgical physician in completing cerebral angiography examination through the operation of experimental instruments or artificial means.

SECONDARY OUTCOMES:
Super-selective Technique Success Rate | at the end of surgery
  Assessing the technical success rate of the surgical physician in performing super-selective catheterization of cerebral vessels through the operation of experimental instruments or artificial means.
Super-selective Catheterization Time for Target Vessels | at the end of surgery
  Calculate and compare the average time taken to perform super-selective catheterization for each target vessel during each surgical procedure.
DSA Fluoroscopy Time | at the end of surgery
  Record and compare the duration of fluoroscopy during DSA for each surgical procedure.
Surgical Time | at the end of surgery
  Record and compare the duration of each surgical procedure.
Primary Operator Radiation Absorbed Dose | at the end of surgery
  Record and compare the absorbed dose of ionizing radiation received by the primary operator during each surgical procedure.
Instrument Performance Evaluation | at the end of surgery
  The surgical physician fills out a form after the surgery to subjectively evaluate the performance of the experimental instruments during the angiographic examination procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai City, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Xu H, Sun J, Chen WH, Zhang Y, Chen M, Yi T, Wu YM, Cheng G, Guo J, Yang P, Guo S, Liu J. Safety and efficacy of cerebral robot assisted angiography: randomized comparison of robotic versus manual procedures. J Neurointerv Surg. 2025 Jul 9:jnis-2025-023412. doi: 10.1136/jnis-2025-023412. Online ahead of print. PMID 40633938